CLINICAL TRIAL: NCT05808803
Title: A Single-center, Retrospective Cohort Study of Aberrant Myeloid Lineage Differentiation in HIV/AIDS Patients
Brief Title: Aberrant Myeloid Lineage Differentiation in HIV/AIDS Patients
Status: Completed | Type: Observational
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 05
Record Dates: First submitted 2023-02-10; First posted 2023-04-11 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-01

CONDITIONS: HIV Infections; Leukemia
MeSH Terms: conditions — HIV Infections; Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV without leukemia
- HIV leukemia

SUMMARY:
The investigators included 782 HIV-infected patients from January 2016 to October 2020 Zhongnan Hospital of Wuhan University, whose AIDS diagnosis criteria met the "AIDS Diagnosis and Treatment Guide (2018 edition)" of Chinese Medical Association.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infection

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators included 782 HIV-infected patients from January 2016 to October 2020 Zhongnan Hospital of Wuhan University, whose AIDS diagnosis criteria met the "AIDS Diagnosis and Treatment Guide (2018 edition)" of Chinese Medical Association. There were 647 male patients and 135 female patients, aged 14-78 years, with an average age of 43 years.
Sampling Method: Non-Probability Sample
Enrollment: 782 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
The proportion of granulocytes and granulocyte/macrophage progenitors in myelogram of HIV/AIDS patients | 2020
  Flow cytometric immunophenotyping of an EDTA-anticoagulated BM aspirate specimen was performed. A standard BM assay with erythrocyte cell lysis was used for all BM aspirate specimens. Flow cytometric analysis was conducted using a FACS Canto II flow cytometer (Becton Dickinson, Sunnyvale, CA, USA).

SECONDARY OUTCOMES:
Neutrophil counts in peripheral blood of HIV/AIDS patients | 2020
  Blood samples were drawn from patients undergoing routine diagnostic blood analysis at our institute by sterile venipuncture into tubes containing 5.4 mg of K2EDTA and analyzed by the automated hematology analyzer.